CLINICAL TRIAL: NCT02737410
Title: Resilience in Irritable Bowel Syndrome and Gut-focused Hypnotherapy: Longitudinal Study With Hypnotherapy Patients and Cross Sectional Control Group
Brief Title: Resilience in Irritable Bowel Syndrome and Gut-focused Hypnotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gabriele Moser, Professor, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 1488/2012
Record Dates: First submitted 2016-01-20; First posted 2016-04-13 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Irritable Bowel Syndrome
Keywords: Resilience; Coping; Psychosomatic; Hypnosis; Construct Validation
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Active Comparator): Treatment group obtaining Gut-directed Hypnotherapy
  Interventions: Behavioral: Gut-directed Hypnotherapy
- Control (No Intervention): Control group

INTERVENTIONS:
Behavioral: Gut-directed Hypnotherapy — The GHT protocol used was the Manchester protocol of GHT and consisted of 10 weekly sessions (45 min), with six patients per group over a treatment period of 12 weeks. GHT was performed at the University Hospital by two experienced physicians trained in Manchester (UK).
  Other Names: Gut-focused Hypnotherapy
  Arms: Treatment

SUMMARY:
Background:

Resilience refers to a class of variables highly relevant for wellbeing and coping with stress, trauma, and chronic adversity. Despite its significance for health, resilience is hardly examined empirically and suffers from poor conceptual integration. Irritable bowel syndrome (IBS) is a functional disorder with altered psychological stress reactivity and brain-gut-microbiota axis, which causes high chronic strain. Gut-focused hypnotherapy (GHT) is a standardized treatment for IBS targeting at resilience. An increase of resilience by GHT has been hypothesized but requires further investigation.

Aims of the study were construct validation and development of an integrational measure of different resilience domains by dimensional reduction, and investigation of change in resilience in IBS patients by GHT.

N=74 Gastroenterology outpatients with Irritable Bowel Syndrome (Rome III criteria) were examined in 7 resilience domains, quality of life, psychological distress and symptom severity. n=53 of these participate in 7 to 10 Gut-directed Hypnotherapy group sessions (Manchester protocol). Post-treatment examinations were performed 10 months after last GHT session.

DETAILED DESCRIPTION:
Aims of this study were, to measure detailed factors of resilience by adequate psychological instruments in a sample of Irritable Bowel Syndrome (IBS) patients and to investigate whether they are facets of the same underlying construct. To calculate a composite measure of resilience based on obtained insights concerning the structure of resilience. To test the hypothesis of a positive relation between resilience and response to therapy. And finally, to investigate differences between patients untreated or treated with Gut-directed Hypnotherapy in groups cross-sectionally and longitudinally, to test the hypothesis of a presumed increase in resilience (using the composite score) with changes in IBS symptoms, quality of life and psychological distress in parallel.

Study location and recruitment:

N=74 Irritable bowel syndrome patients (diagnosed according to Rome III criteria) aged between 18 and 70 and refractory to other therapies were recruited at the Specialized outpatient-clinic for Psychosomatics at the Division of Gastroenterology and Hepatology, Department for Internal Medicine III, University Hospital of Vienna. Antidepressants or anxiolytics and/or ongoing psychotherapy were allowed since severe comorbid psychological problems are a common problem in IBS patients. The study protocol was approved by the ethics committee of the Medical University of Vienna (ID: 1488/2012). Informed consent in writing was given by each participant.

Study Design and Treatment:

Cross-sectional comparisons were performed with data of n = 37 GHT treated and n = 37 untreated patients (control group) post GHT. This data were pooled for dimensional reduction of resilience domains. Resilience and IBS severity data from the treatment group were assessed post GHT; psychological distress and quality of life were assessed pre and post GHT. A fraction of n = 16 of the untreated patients (former control group) subsequently also received GHT treatment. Pre and post GHT data of these patients were collected and then used for longitudinal comparisons, along with the pre and post GHT data on psychological distress and quality of life of the primary treatment group. In total, N= 74 patients were examined, in total 53 (= 37 + 16) of which underwent GHT. Post treatment examinations were performed 10 months after last GHT session. The GHT protocol used was the Manchester protocol of GHT and consisted of 10 weekly sessions (45 min), with six patients per group over a treatment period of 12 weeks. GHT was performed at the University Hospital by two experienced physicians trained in Manchester (UK).

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of IBS (Rome-III-criteria)
* Indication of GHT because of no adequate relief of IBS symptoms and no improvement of disease-related quality of life through other IBS therapies

Exclusion Criteria:

* pregnancy, mental retardation
* insufficient knowledge of German
* transit time from home to hospital longer than one hour

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-06; Primary Completion 2014-06 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Resilience assessed using the Connor-Davidson Resilience Scale | 1 year
  10-item Connor-Davidson Resilience Scale, with higher values indicating higher resilience.
Self-efficacy assessed by the Skala zur allgemeinen Selbstwirksamkeitserwartung | 1 year
  Skala zur allgemeinen Selbstwirksamkeitserwartung (SWE) is a german questionnaire to assess self-efficacy. Higher values mean higher self-efficacy.
Humor assessed by the State-Trait Cheerfulness Inventory | 1 year
  State-Trait Cheerfulness Inventory, german version (STCI); higher values indicate higher predisposition to experience positive emotion by humor.
Social support assessed by the Fragebogen zur Sozialen Unterstützung | 1 year
  Fragebogen zur Sozialen Unterstützung (F-SozU), a german Questionnaire assessing perceived social support, with higher values indicating higher perceived support.
Emotion regulation assessed by the Cognitive Emotion Regulation Questionnaire | 1 year
  Cognitive Emotion Regulation Questionnaire (CERQ), german version; assessing adaptive and dysfunctional cognitive reactions to aversive events. Higher values represent higher occurence of respective behaviours.
Neuroticism assessed by the Big Five Inventory | 1 year
  Big Five Inventory, german short form (BFI-K), for assessment of neuroticism. Higher values indicate higher neuroticism.

SECONDARY OUTCOMES:
Psychological distress assessed by the Hospital Anxiety and Depression Scale | 1 year
  The Hospital Anxiety and Depression Scale (German version, HADS-D) is an instrument for screening anxiety and depression in primarily somatic ill patients. Higher values indicate more distress.
Quality of life assessed by visual analogue scales | 1 year
  Quality of life was assessed via single visual analogue scales (VAS). Higher values represent higher wellbeing.
Symptom severity assessed by the Irritable Bowel Syndrome - Severity Scoring System | 1 year
  The Irritable Bowel Syndrome - Severity Scoring System (IBS-SSS) is a questionnaire for clinical assessment of IBS symptom burden and severity. Higher values indicate higher symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriele Moser, Professor, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Yes
via www.figshare.com